CLINICAL TRIAL: NCT05546138
Title: Characterization and Prediction of Early Onset Diabetic Peripheral Neuropathy (NeuroPredict)
Brief Title: Characterization and Prediction of Early Onset Diabetic Peripheral Neuropathy
Acronym: NeuroPredict
Status: Recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other); University of Aarhus (Other)
Responsible Party: Principal Investigator, Johan Bovbjerg Røikjer, Primary Investigator, Aalborg University Hospital
Other Study IDs: N-20220013
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Neuropathy, Diabetic; Small Nerve Fiber Neuropathy; Type 1 Diabetes
Keywords: Diabetic neuropathy, Early detection, Clinical Endpoints, Prediction, Risk stratification
MeSH Terms: conditions — Diabetic Neuropathies; Small Fiber Neuropathy; Diabetes Mellitus, Type 1 | interventions — Magnetic Resonance Imaging; Diffusion Tensor Imaging; Nerve Conduction Studies; Surveys and Questionnaires; diazonaphthalenedisulfonic acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 1 diabetes without known peripheral neuropathy: People with type 1 diabetes without known peripheral neuropathy with "limited" diabetes duration
  Interventions: Diagnostic Test: Skin biopsies with quantification of intra-epidermal nerve fibre density; Diagnostic Test: Perception Threshold Tracking; Diagnostic Test: Thermal perception thresholds; Diagnostic Test: Corneal confocal Microscopy; Diagnostic Test: MRI; Diagnostic Test: Nerve conduction studies; Other: Composite scores and questionnaires

INTERVENTIONS:
Diagnostic Test: Skin biopsies with quantification of intra-epidermal nerve fibre density — Skin biopsy
  Other Names: PGP9.5, antibodies for subsets of ion-channels ect
Diagnostic Test: Perception Threshold Tracking — Transcutaneous stimulation of large and small nerve fibres using weak electrical currents
  Other Names: PTT
Diagnostic Test: Thermal perception thresholds — Heat and cold perception thresholds
  Other Names: Quantitative Sensory Testing
Diagnostic Test: Corneal confocal Microscopy — Corneal nerve fibre density, corneal nerve fibre length, corneal nerve branch density
  Other Names: CCM
Diagnostic Test: MRI — Functional and structural MRI pictures of peripheral nerves and CNS
  Other Names: fMRI, DTI, neurography
Diagnostic Test: Nerve conduction studies — Nerve conduction and amplitude of Sural nerve
  Other Names: NC-STAT DPNCheck
Other: Composite scores and questionnaires — Composite scores and questionnaires
  Other Names: DN4, MNSI, NDS, NAFF

SUMMARY:
Predicting early onset neuropathy in people with type 1 diabetes

DETAILED DESCRIPTION:
Background

Diabetic peripheral neuropathy is the most common complication to diabetes mellitus affecting as much as 50% of the population with diabetes. Symmetrical sensory neuropathy is by far the most common pattern, which often progress slowly over many years, although some individuals experience faster and more severe courses. Despite the frequent occurrence, the causes of diabetic peripheral neuropathy are largely unknown, which is reflected in the fact that no disease-modifying treatments are available for preventing, treating or even halting the progression of the disease. The consequences can be dire, as neuropathy frequently leads to foot ulcers, amputations or intolerable neuropathic pain in the lower extremities. Sensory loss may go completely undetected in diabetes, as there often are literally no symptoms. For many individuals, the development of diabetic peripheral neuropathy can therefore proceed completely unnoticed, making regular screening the most important tool for diagnosing the condition. Unfortunately, unlike nephropathy or retinopathy, diabetic peripheral neuropathy is not easily screened for, as the condition lacks reliable markers for early- or progressing disease. Therefore, screening for diabetic peripheral neuropathy currently revolves around diagnosing loss of protective sensation, judged by the inability to feel vibration or light touch. However, in their most recent guidelines, the American Diabetes Association has included screening for small fibre neuropathy using either the cold- and heat perception thresholds or pinprick as a clinical standard. Although this acknowledgement of the importance of assessing not only large- but also small nerve fibres is a huge step towards early detection of diabetic peripheral neuropathy, the overriding issue of insensitive, unreproducible, and inaccurate bedside tests for small nerve fibres remains. While cold- and heat perception and pinprick sensation are indeed mediated by small nerve fibres, the sensitivity of these methods, outside of extreme standardization only achievable in dedicated neuropathy research-centres, remain poor and not usable on an individual level. This lack of sensitivity has also become apparent in several large clinical trials, where the methods have continuously failed as robust clinical endpoints. Due to this, the hunt for a sensitive and reproducible method for adequate assessment of the small nerve fibres have begun. Amongst several interesting methods, two have gained particular interest (corneal confocal microscopy and skin biopsies with quantification of intra-epidermal nerve fibre density), due to their diverse strengths, although clinical application is currently limited to a few specialized sites. Furthermore, both methods suffer several inherent issues including that fact that they only provide information about the structure of the nerves and not the function.

In this study, we will therefore combine established gold standards for early detection of structural changes to small nerve fibres in diabetic peripheral neuropathy with cutting-edge, experimental techniques for measuring the function of the same nerve fibres. Furthermore, we will also evaluate several advanced technologies as an alternative to the current clinical standard for large fibre evaluation (biothesiometry).

Study objectives

* To establish a prospective cohort for long-term follow-up for early detection of the development of diabetic peripheral neuropathy
* To evaluate alternative methods for screening for diabetic peripheral neuropathy in a clinical setting
* To evaluate measurements of small nerve fibre function against methods for small nerve fibre structure

Methods

A prospective, long-term, follow-up, cohort study running from 01.04.2022-31.12.2029. The study will consist of two different, yet aligned, sub-studies:

1. An observational, cohort study consisting of a random sample of up to 1,000 persons with diabetes (any type) and neuropathy at any stage, entering the outpatient clinic at Steno Diabetes Center North Denmark/Department of Endocrinology, Aalborg University Hospital.
2. A smaller, observational, cohort study consists of 100-200 persons with type 1 diabetes and no clinically detectable neuropathy.

The first study will aim to evaluate alternative screening methods to be used in clinical practice, while it will also be used to identify persons eligible to participate in the second study.

The second study will aim to preform deep-sensory phenotyping of people without established diabetic peripheral neuropathy using methods evaluating both structure and function of small nerve fibers. The cohort will be followed from inclusion and evaluated once yearly to see if they are progressing. Ultimately, this cohort will be used to retrospectively evaluate, if any, or a combination of, the used experimental methodology can predict, who develops diabetic peripheral neuropathy, and who doesn't.

Participants from either of the two studies will be informed about the trial and their expected outcomes both written and vocally. Participants will follow their usual clinical control for diabetes and complication-screening (including usual foot care and neuropathy screening), and the enhanced screening performed in this study will therefore be an addition to clinical standard. No interventions will be made.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-80 years
* Diagnosed with diabetes (of any type)
* No clinically established diabetic peripheral neuropathy at inclusion

Exclusion Criteria:

* Alcohol or drug abuse within the last year (prior to inclusion)
* Chemotherapy (prior or within study period) or experimental medicine
* Severe vitamin deficiencies
* Inability to understand or comply with the examinations
* Planned or likely discontinuation of care at Aalborg University Hospital
* Known hematologic disorders resulting in a markedly reduced ability to stop small bleedings
* Severe limb ischemia
* Active diabetic foot ulcers
* Previous amputations
* Severe skin diseases or diseases known to cause neural damage
* Pregnancy at inclusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Type 1 diabetes without established neuropathy with planned continuity of care at Steno Diabetes Center North Denmark, Aalborg
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Prediction of early onset neuropathy | 1,3,5,7,9 years
  Retrospective evaluation of the predictive power for each of the diagnostic tests
Comparison of Perception Threshold Tracking (PTT) and skin biopsies | 1-2 years
  Sensitivity, specificity, PPV, NPV of PTT compared to skin biopsies
Progression and regression of neuropathy | 1-9 years
  Description of the natural history of the development of neuropathy

SECONDARY OUTCOMES:
Development and testing of single-use electrode for PTT | 5 years
  As title states
Development and testing of new pulse shapes for PTT | 5 years
  As title states
Correlation between central and peripheral measurements | 1-5 years
  MRI-scans vs peripheral measurements

OTHER OUTCOMES:
Stability of skin biopsies over time | 9 years
  Repeated analysis of intra-epidermal nerve fibre density in skin biopsies frozen several years
fMRI as a marker for progression of neuropathy | 9 years
  as title states

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vestergaard, PhD, Study Chair — Steno Diabetes Center North Denmark; Johan M Røikjer, PhD, Principal Investigator — Steno Diabetes Center North Denmark
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Steno Diabetes Center North Denmark — https://stenodiabetescenter.rn.dk/